CLINICAL TRIAL: NCT02100358
Title: Accuracy of Functional MRC With Gadoxetate Disodium in the Diagnosis of Acute Cholecystitis: Comparison With Hepatobiliary Scintigraphy
Brief Title: Functional MRC With Eovist for Acute Cholecystitis
Acronym: MRC
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 403462
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute cholecystitis: acute cholecystitis

SUMMARY:
Functional magnetic resonance cholangiography (fMRC) with gadoxetate disodium (Eovist) is an accurate method of diagnosing acute cholecystitis.

DETAILED DESCRIPTION:
Primary Objective:

To determine the accuracy of fMRC in evaluating patients with suspected cholecystitis.

Secondary Objective:

To compare the results of fMRC with conventional hepatobiliary scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Symptoms of right upper quadrant pain with ambiguous US (and/or CT) findings
* Standard of care nuclear medicine hepatobiliary scan to rule out acute cholecystitis -

Exclusion Criteria:

* Scheduled for emergent surgery, or is otherwise determined by the Investigator that the subject is clinically unsuitable for the study
* Glomerular filtration rate (GFR) below 60 mL/min/1.73m2
* Total bilirubin above 3.0 mg/dL
* Inability to provide informed consent (altered or diminished mental status)
* Allergic to morphine
* Known or suspected hypersensitivity to gadolinium-based agents
* The standard MRI contraindications apply, including but not limited to: having a pacemaker or other implanted electronic device, metal foreign bodies within the eye, aneurysm clips, heart valve prosthesis, vascular stents, coils, intrauterine devices (IUDs), penile implants, inferior vena cava (IVC) filters, gunshot wounds with retained bullet fragments.
* Pregnant or breast-feeding -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have recently (within 12 hours) undergone a clinically-indicated nuclear medicine hepatobiliary scan not involving sedation or anesthesia for suspected acute cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of positive cases of acute cholecystitis | 2 years
  The primary outcome measure is the number of positive cases of acute cholecystitis on functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Corwin, MD, Principal Investigator — Assistant Professor
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States